CLINICAL TRIAL: NCT05779501
Title: Testing the Efficacy of an Internet-delivered Strengths Use Intervention in Organizations A Waiting-list Randomized Trial
Brief Title: Efficacy of Internet-delivered Strengths Use Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West University of Timisoara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: MEGSIS S3 RCT
Record Dates: First submitted 2023-02-27; First posted 2023-03-22 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-02

CONDITIONS: Mental Health Wellness; Professional Burnout
MeSH Terms: conditions — Burnout, Professional | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: Two-armed randomized trial with waiting-list control and pre-, mid-, and post-intervention measurements.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The experimental arm will receive the online strengths use intervention program over a period of 4 weeks, through an LMS software solution.
  Interventions: Behavioral: Internet-delivered strengths use intervention
- Waiting-list control group (Other): The waiting-list control arm will receive the same intervention immediately after the intervention group finishes and will have filled in the post-test outcomes measures.
  Interventions: Behavioral: Waiting-list

INTERVENTIONS:
Behavioral: Internet-delivered strengths use intervention — The online strengths use intervention program follows the theorized five stages of strengths use interventions: (1) preparation and commitment, (2) identification, (3) integration, (4) action, and (5) evaluation. To increase participant engagement and motivation, gamification components are embedded in several stages.
  The intervention was previously tested through a feasibility and acceptability trial (NCT05474807).
  The entire intervention will be delivered online via an LMS software solution.
  Arms: Intervention group
Behavioral: Waiting-list — The waiting-list arm will serve as the control group, filling in only the outcome measure at the same time as the intervention group participants.
  After the intervention group finishes participating in the intervention, the waiting-list participants will benefit from the same internet-delivered strengths use program.
  Arms: Waiting-list control group

SUMMARY:
The aim of the study will be to test the efficacy of a novel online-delivered gamification-based intervention for the identification, development, and use of strengths in the workplace. The program will be addressed to young employees and will have the aim of boosting their well-being and performance.

ELIGIBILITY:
Inclusion Criteria:

* Not other than the age of the participants.

Exclusion Criteria:

* Lack of internet access during the period of the implementation of the program (prescreened during enrolment).

Controlled variables:

* Participants levels of work engagement and work experience will be controlled for by stratified randomization. For each of the two factors we will created three strata (low level: lowest - 33rd percentile; moderate level: 34th - 66th percentile; high level: 67th percentile - highest), and the randomization will be applied for each stratum.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 167 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Work engagement | Change from baseline to mid-intervention and post-intervention (approximately 3 weeks and 6 weeks).
  Work engagement will be measured with the Utrecht Work Engagement Scale (UWES-9). It has 9 items that form three dimensions, each with 3 items: vigor (e.g., "At my work, I feel bursting with energy"), dedication (e.g., "I am enthusiastic about my job"), and absorption (e.g., "I am immersed in my work"). This measure uses a 7-point scale (0 =never, 6 = always). Higher scores represent higher work engagement.
Psychological capital (PsyCap) | Change from baseline to mid-intervention and post-intervention (approximately 3 weeks and 6 weeks).
  Psychological capital will be measured with the 12-item Psychological Capital Questionnaire. It has four subscales: hope ("At the moment, I feel quite fulfilled at work."), self-efficacy ("I feel confident presenting information to a group of colleagues."), resilience ("Usually, at work, I easily get over the stressful aspects."), and optimism ("I am optimistic about what will happen to me in the future regarding my job."). All 12-item are reported on a 6-point Likert scale (1 = strongly disagree, 6 = strongly agree). Higher scores represent higher PsyCap.
Strengths use | Change from baseline to mid-intervention and post-intervention (approximately 3 weeks and 6 weeks).
  The Strengths Use subscale from the Strengths Use and Deficit Correction questionnaire (SUDCO). I has 6 items, rated on a 0 (almost never) to 6 (almost always) scale. A sample item is "I seek opportunities to do my work in a manner that best suits my strong points". Higher scores represent higher levels of strengths use.
Strengths identification, use and development | Change from baseline to mid-intervention and post-intervention (approximately 3 weeks and 6 weeks).
  A set of 18 items, rated on a 0 (almost never) to 6 (almost always) scale, was developed by the team of experts involved in this study. Higher scores represent higher levels of strengths use, identification, and development.

SECONDARY OUTCOMES:
Burnout | Change from baseline to post-intervention (approximately 6 weeks).
  Burnout will be assessed with the 12-item Burnout Assessment Tool (BAT). This questionnaire has four subscales: exhaustion (3 items; "At work, I feel mentally exhausted."), emotional impairment (3 items; "At work, I feel unable to control my emotions."), cognitive impairment (3 items; "At work, I have trouble staying focused.") and mental distance (3 items; "I struggle to find any enthusiasm for my work."). All items are scored on a 5-point scale ranging from 1(never) to 5 (always). Higher scores represent elevated symptoms of burnout.
Job satisfaction | Change from baseline to post-intervention (approximately 6 weeks).
  Job satisfaction will be measured with the Michigan Organizational Assessment Questionnaire. The scale has three items with a response on a 7-point Likert scale (1 = total disagreement, 7 = total agreement). A sample item reads: "In general, I like working here.". Higher scores represent higher job satisfaction.
Job performance | Change from baseline to post-intervention (approximately 6 weeks).
  Job performance will be assessed with a 7-item scale. Response options range on a Likert scale from 1 (strongly disagree) to 5 (strongly agree). A sample item is "I adequately complete my assigned duties.". Higher scores represent higher performance.
Employability | Change from baseline to post-intervention (approximately 6 weeks).
  Employability will be measured with the four-item Perceived Employability Scale. Each item is rated on a 5-point Likert scale (1 = totally disagree; 5 = totally agree). Higher scores represent higher levels of employability.

OTHER OUTCOMES:
Life satisfaction | Change from baseline to post-intervention (approximately 6 weeks).
  Life satisfaction will be measured with the five items of the Satisfaction with Life Scale. All answers are reported on a 7-point Likert scale (1 = totally disagree; 7 = totally agree); one item example being, "I am satisfied with my life". Higher scores represent higher satisfaction with life.
Satisfaction with the intervention | At study completion (post-intervention), an average of 6 weeks.
  Satisfaction with the intervention will be measured using 38 items. A higher score means a better outcome (increased satisfaction with the intervention).
Satisfaction with the intervention | At study completion (post-intervention), an average of 6 weeks.
  7 open-ended questions exploring participants' subjective experience with the intervention program.

CONTACTS AND LOCATIONS:
Locations (1):
- West University of Timisoara, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Camman, C., Fichman, M., Jenkins, D., & Klesh, J. (1979). The Michigan Organizational Assessment Questionnaire(University of Michigan, Ann Arbor, Michigan).
- [Background] Luthans, F. L., Avolio, B. J., & Avey, J. A. (2007). Psychological Capital Questionnaire (PsyCap) [Database record]. APAPsycTests. https://doi.org/10.1037/t06483-000
- [Background] Schaufeli, W. B., Bakker, A. B., & Salanova, M. (2006). The measurement of work engagement with a short questionnaire: Across-national study. Educational and psychological measurement, 66(4), 701-716.https://doi.org/10.1177/0013164405282471
- [Background] Schaufeli WB, Desart S, De Witte H. Burnout Assessment Tool (BAT)-Development, Validity, and Reliability. Int J Environ Res Public Health. 2020 Dec 18;17(24):9495. doi: 10.3390/ijerph17249495. PMID 33352940
- [Background] Tulbure BT, Rusu A, Sava FA, Salagean N, Farchione TJ. A Web-Based Transdiagnostic Intervention for Affective and Mood Disorders: Randomized Controlled Trial. JMIR Ment Health. 2018 May 24;5(2):e36. doi: 10.2196/mental.8901. PMID 29798831
- [Background] Van Woerkom, M., Mostert, K., Els, C., Bakker, A. B., De Beer, L., & Rothmann Jr, S. (2016). Strengths use and deficit correction in organizations: Development and validation of a questionnaire. European Journal of Work and Organizational Psychology, 25(6), 960-975. https://doi.org/10.1080/1359432X.2016.1193010
- [Background] Watson D, Clark LA. Negative affectivity: the disposition to experience aversive emotional states. Psychol Bull. 1984 Nov;96(3):465-90. No abstract available. PMID 6393179
- [Background] Williams, L. J., & Anderson, S. E. (1991). Job satisfaction and organizational commitment as predictors of organizational citizenship and in-role behaviors. Journal of management, 17(3), 601-617. https://doi.org/10.1177/014920639101700305
- [Background] Miglianico, M., Dubreuil, P., Miquelon, P., Bakker, A. B., & Martin-Krumm, C. (2020). Strength use in the workplace: aliterature review. Journal of Happiness Studies, 21(2), 737-764. https://doi.org/10.1007/s10902-019-00095-w
- [Background] De Witte, H. (1992). Tussen optimisten en teruggetrokkenen. Een empirisch onderzoek naar het psychosociaal profiel vanlangdurig werklozen en deelnemers aan de Weer-Werkactie in Vlaanderen [Between optimists and withdrawns. An empiricalinvestigation of the psychosocial profile of longterm unemployed and participants of the Back-to-Work Program in Flanders].Leuven, Belgium: HIVA